CLINICAL TRIAL: NCT02955251
Title: A Multi-Center, Phase 1, Open-Label, Dose-Escalation Study of ABBV-428, an Immunotherapy in Subjects With Advanced Solid Tumors
Brief Title: A Study of ABBV-428, an Immunotherapy, in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-819; 2016-001461-88 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Cancer; Neoplasm; Advanced solid tumor; Nivolumab; Non-small cell lung cancer (NSCLC); Non-squamous NSCLC; Ovarian cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms | interventions — ABBV-428; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (Experimental): ABBV-428 will be administered at escalating dose levels in 28-day dosing cycles (2 doses per cycle).
  Interventions: Drug: ABBV-428
- Arm A, B, and C (Experimental): Additional participants (with ovarian cancer, NSCLC, etc.) will be enrolled in a dose expansion cohorts that will further evaluate ABBV-428.
  Interventions: Drug: ABBV-428
- Arm D (Experimental): Additional participants with NSCLC will be enrolled in an expansion cohort that will further evaluate ABBV-428 plus nivolumab.
  Interventions: Drug: ABBV-428; Drug: Nivolumab
- Arm 2 (Experimental): ABBV-428 plus nivolumab.
  Interventions: Drug: ABBV-428; Drug: Nivolumab

INTERVENTIONS:
Drug: ABBV-428 — ABBV-428 will be administered by intravenous infusion in 28-day dosing cycles on Day 1 and Day 15.
Drug: Nivolumab — Nivolumab will be administered by intravenous infusion according to approved dose and dosing schedules.
  Other Names: OPDIVO
  Arms: Arm 2; Arm D

SUMMARY:
This is an open-label, Phase I, dose-escalation study to determine the recommended Phase 2 dose (RPTD), maximum tolerated dose (MTD), and evaluate the safety and pharmacokinetic (PK) profile of ABBV-428 when administered as monotherapy or in combination with nivolumab in participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an advanced solid tumor that has progressed on standard therapies known to provide clinical benefit or the participants are intolerant to such therapies.
* Participants have adequate bone marrow, renal, hepatic and coagulation function.
* For all dose expansion arms, participants must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
* Participants in combination therapy cohorts must have an advanced solid tumor where the use of nivolumab is standard therapy.

Exclusion Criteria:

* Active or prior documented autoimmune disease in the last 2 years. Participants with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose (with certain exceptions).
* History of primary immunodeficiency, bone marrow transplantation, chronic lymphocytic leukemia, solid organ transplantation, or previous clinical diagnosis of tuberculosis.
* Confirmed positive test results for human immunodeficiency virus (HIV), or participants with chronic or active hepatitis B or C. Participants who have a history of hepatitis B or C who have undetectable HBV DNA or HCV RNA after anti-viral therapy may be enrolled.
* Prior grade greater than or equal to 3 immune-mediated neurotoxicity or pneumonitis (or any other unresolved or symptomatic adverse event in the last 3 months) while receiving immunotherapy.
* Male participants who are considering fathering a child or donating sperm during the study or for at least 3 or 5 months (for monotherapy and combination therapy participants, respectively) after the last dose of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | First dose of study drug through at least 100 days after end of treatment; up to 2 years after last participants first dose
Recommended Phase 2 Dose (RPTD) of ABBV-428 when administered as monotherapy or in combination with nivolumab | 1 day of study drug administration within the 28-day cycle at the designated cohort dose
  If a maximum tolerated dose (MTD) is reached, the RPTD of ABBV-428 will not be a dose higher than the defined MTD, and will be selected based on the type(s) and occurrence(s) of dose limiting toxicities which occur in addition to the MTD. If a MTD is not reached, then the RPTD will be defined based on the safety and pharmacokinetic data.
Area under the serum concentration-time curve (AUC) of ABBV-428 | Up to 30 days after a 24-month treatment period
Terminal half-life (t1/2) of ABBV-428 | Up to 30 days after a 24-month treatment period
Maximum observed serum concentration (Cmax) of ABBV-428 | Up to 30 days after a 24-month treatment period
Maximum tolerated dose (MTD) of ABBV-428 when administered as monotherapy or in combination with nivolumab | Up to 2 years
  The highest dose level at which less than 2 of 6 participants or less than 33% of (if cohort is expanded beyond 6) participants experience a dose limiting toxicity.
Time to Cmax (Tmax) of ABBV-428 | Up to 30 days after a 24-month treatment period

SECONDARY OUTCOMES:
Duration of Objective Response (DOR) | Up to 30 days after a 24-month of treatment period
  DOR defined as the time from the initial objective response to disease progression or death, whichever occurs first.
Clinical benefit rate (CBR) | Up to 30 days after a 24-month of treatment period
  CBR defined as the proportion of subjects with a confirmed partial response (PR), complete response (CR), or stable disease for at least 24 weeks to the treatment.
Progression-Free Survival (PFS) | Up to 30 days after a 24-month of treatment period
  PFS time is defined as the time from the first dose of ABBV-428 to disease progression or death, whichever occurs first
Objective Response Rate (ORR) | Up to 30 days after a 24-month of treatment period
  ORR is defined as the proportion of subjects with a confirmed partial or complete response to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (15):
- United States (7):
  - HonorHealth Research Institute - Pima /ID# 155461, Scottsdale, Arizona
  - UC Davis Comprehensive Cancer Center - Main /ID# 154439, Sacramento, California
  - University of Chicago /ID# 154440, Chicago, Illinois
  - Fox Chase Cancer Center /ID# 170665, Philadelphia, Pennsylvania
  - Greenville Hospital System /ID# 154437, Greenville, South Carolina
  - MD Anderson Cancer Center at Texas Medical Center /ID# 154441, Houston, Texas
  - South Texas Accelerated Research Therapeutics /ID# 154442, San Antonio, Texas
- Australia (2):
  - Chris O'Brien Lifehouse /ID# 163131, Camperdown, New South Wales
  - Northern Cancer Institute /ID# 163132, St Leonards, New South Wales
- France (5):
  - Institut Bergonie /ID# 202391, Bordeaux, Gironde
  - Hopital de la Timone /ID# 162256, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Leon Berard /ID# 168072, Lyon, Rhone
  - Institut Curie /ID# 162258, Paris, Île-de-France Region
  - Gustave Roussy /ID# 162257, Villejuif, Île-de-France Region
- National Taiwan Univ Hosp /ID# 169034, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luke JJ, Barlesi F, Chung K, Tolcher AW, Kelly K, Hollebecque A, Le Tourneau C, Subbiah V, Tsai F, Kao S, Cassier PA, Khasraw M, Kindler HL, Fang H, Fan F, Allaire K, Patel M, Ye S, Chao DT, Henner WR, Hayflick JS, McDevitt MA, Fong L. Phase I study of ABBV-428, a mesothelin-CD40 bispecific, in patients with advanced solid tumors. J Immunother Cancer. 2021 Feb;9(2):e002015. doi: 10.1136/jitc-2020-002015. PMID 33608377